CLINICAL TRIAL: NCT04155502
Title: Using Social Media to Deliver HIV Self-Testing Kits and Link to Online PrEP Services
Acronym: CTN-0083
Status: Completed | Type: Observational
Sponsor: Lisa A. Marsch (Other)
Collaborators: National Drug Abuse Treatment Clinical Trials Network (Network); University of California, Los Angeles (Other); Dartmouth College (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Lisa A. Marsch, Professor, Dartmouth-Hitchcock Medical Center
Organization: Dartmouth-Hitchcock Medical Center (Other)
Other Study IDs: CTN-0083, STUDY00031899; UG1DA040309 (NIH)
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: HIV Infections
Keywords: HIV; Pre-exposure prophylaxis; Social media; Online advertising
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Social media sites.: These participants will be recruited from advertisements posted on social media websites. Participants who complete the baseline assessment will receive a code to order a free HIV self-test kit. Participants will be asked to complete two online follow-up questionnaires at 14-days and 60-days post-baseline. These questionnaires will ask questions related to HIV self-test kit use and PrEP uptake.
- Informational sites: These participants will be recruited from advertisements posted on informational websites. Participants who complete the baseline assessment will receive a code to order a free HIV self-test kit. Participants will be asked to complete two online follow-up questionnaires at 14-days and 60-days post-baseline. These questionnaires will ask questions related to HIV self-test kit use and PrEP uptake.
- Dating applications: These participants will be recruited from advertisements posted on dating applications. Participants who complete the baseline assessment will receive a code to order a free HIV self-test kit. Participants will be asked to complete two online follow-up questionnaires at 14-days and 60-days post-baseline. These questionnaires will ask questions related to HIV self-test kit use and PrEP uptake.

SUMMARY:
The primary objective of this study is to compare the relative effectiveness of three web-based platforms: social media sites (e.g., Facebook), dating applications [apps] (e.g., Grindr), and informational sites (e.g., Google) to promote self-testing of Human Immunodeficiency Virus (HIV) infection among men who have sex with men (MSM) who are at increased risk of HIV exposure and/or infection. In addition, we will measure Pre-Exposure Prophylaxis (PrEP) uptake and evaluate the degree to which substance use and, separately, the participant's intention to test affect HIV self-testing and PrEP uptake. Through this research, we will also examine how participants' social media use, attitudes on HIV testing, perceptions of sexual risk behavior, medical mistrust, and stigma impact HIV testing and PrEP uptake.

DETAILED DESCRIPTION:
Culturally appropriate advertisements (designed specifically for the study population and advertisement method) for promoting HIV testing and PrEP uptake will be created by the study team. These advertisements will be placed on social media sites (Facebook, Instagram, Twitter), informational sites (Google, Bing, Yahoo) and dating apps (Grindr, Hornet, Jack'd) in the form of blast advertisements ("ads"). The advertisements will display on specific days and times (e.g., high traffic utilization) in the geographical locations selected for participation in the study.

Upon clicking the ad, users will land on the study informational page on Qualtrics, where they will receive information about the study, undergo eligibility screening and, if eligible, electronically sign the informed consent. Participants will receive information about HIV testing and PrEP and will be asked to complete the baseline assessment and order their HIV home self-test kit.

Participants will be followed up at two intervals after the baseline assessment. The first will occur 14 days post-baseline, where participants will be asked about their test use and may be asked if they visited a PrEP provider and/or if they started PrEP and about PrEP opinions and facilitators and barriers. If they tested positive for HIV on the home self-test kit, they will be asked whether they have visited an HIV treatment provider. Participants will be asked to upload a picture of their test result for validation on the secure Qualtrics server during the 14-day follow-up assessment. Photographs will be interpreted by the study team and the result will be entered into the study database; photographs will then be deleted.

At the 60-day follow-up, all participants will be asked to respond to study evaluation questions. Additionally, participants may respond to a subset of the questions that is the same as the 14-day follow-up, based on their responses on the first follow-up survey. Those who reported that they received a negative HIV self-test result and started PrEP at the 14-day follow-up will not be asked to answer these questions at the 60-day follow-up. Participants who either did not take the HIV test or did not start PrEP by the 14-day follow-up may be asked about PrEP facilitators and barriers, their self-test use, if they visited a PrEP provider, whether they started PrEP, and if applicable, whether they have visited an HIV treatment provider, depending on their responses during the 14-day follow-up. Participants will be asked to upload a picture of their test result (unless provided at the 14-day follow-up) for validation on the secure Qualtrics server during the 60-day follow-up assessment. Photographs will be interpreted by the study team and the result will be entered into the study database; photographs will then be deleted.

Participants who report a preliminary positive, invalid, or indeterminate result on the HIV home self-test kit will be referred to local brick-and-mortar clinics for additional services and asked to continue participating in follow-up assessments. Regardless of their result, all participants will be offered information on HIV and STD prevention, and locations of clinics and PrEP providers near them.

Data will be collected both indirectly from each website's metrics and directly from the online questionnaires that the participants will complete.

ELIGIBILITY:
Inclusion Criteria:

1. Have clicked on one of the study-specific advertisements posted on the platforms/ websites;
2. Have been biologically born male (cis-gender man), per participant self-report;
3. Report condomless anal intercourse and more than one male sex partner in the 90 days prior to the date of the screening questionnaire;
4. Be between the ages of 18-30 years old, inclusive;
5. Self-identify as Latino and/or Black/African American;
6. Not currently on PrEP and haven't taken PrEP in the last six months prior to the date of the screening questionnaire (per participant self-report);
7. Have not tested for HIV in the last 3 months prior to the date of the screening questionnaire (per participant self-report);
8. Have a Facebook account (for identity validation to reduce duplicate attempts at enrollment); and
9. Be willing to provide contact information (phone number, email) to the study team.

Exclusion Criteria:

1. Are unwilling or unable to provide informed consent.
2. Are unwilling to provide contact information (phone number, email address).
3. Report having a preliminary positive or positive HIV result in a test completed less than 30 days prior to the date of screening or report being currently under treatment for HIV infection.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This study will be recruiting individuals who were biologically born male and identify as men.
Study Population: This study is recruiting men who have sex with men who actively use social media sites, dating apps, or informational sites.
Sampling Method: Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2020-09-20 (Actual); Study Completion 2020-09-25 (Actual)

PRIMARY OUTCOMES:
Self-test kit orders | 60 days
  The daily rate (number of study participants per day) requesting an HIV home self-test kit by promotional platform (social media, informational, dating sites).

SECONDARY OUTCOMES:
Self-test kit use | 60 days
  The number of participants who used the study-provided HIV home self-test kit by 60-day follow-up will be collected via self-report at the time of follow-up (either 14-day or 60-day).

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey D. Klausner, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA David Geffen School of Medicine, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified dataset will be posted on the funder's datashare website. This plan will be described in the study's consent procedures.
Supporting Information: Study Protocol
Time Frame: Data will be provided to NIDA CCTN-designated parties for posting on the NIDA Data Share website after completion of the study and data lock.
Access Criteria: Per the NIDA Data Share 2.0 website:
  "Prior to downloading any study data, the user will be prompted to complete a registration agreement for data use. Users will have to register a name and valid e-mail address in order to download data and to accept their responsibility for using data in accordance with the NIDA Data Share Agreement."
URL: https://datashare.nida.nih.gov/

REFERENCES:
- [Derived] Stafylis C, Vavala G, Wang Q, McLeman B, Lemley SM, Young SD, Xie H, Matthews AG, Oden N, Revoredo L, Shmueli-Blumberg D, Hichborn EG, McKelle E, Moran LM, Jacobs P, Marsch LA, Klausner JD. Relative Effectiveness of Social Media, Dating Apps, and Information Search Sites in Promoting HIV Self-testing: Observational Cohort Study. JMIR Form Res. 2022 Sep 23;6(9):e35648. doi: 10.2196/35648. PMID 36149729
- [Derived] Lemley SM, Klausner JD, Young SD, Stafylis C, Mulatya C, Oden N, Xie H, Revoredo L, Shmueli-Blumberg D, Hichborn E, McKelle E, Moran L, Jacobs P, Marsch LA. Comparing Web-Based Platforms for Promoting HIV Self-Testing and Pre-Exposure Prophylaxis Uptake in High-Risk Men Who Have Sex With Men: Protocol for a Longitudinal Cohort Study. JMIR Res Protoc. 2020 Oct 19;9(10):e20417. doi: 10.2196/20417. PMID 33074164